CLINICAL TRIAL: NCT04586569
Title: A Single Blinded Randomized Controlled Trial Testing the Efficacy of a Pediatric Interactive Relational Agent vs. Standard Preoperative Education
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Boston Children's Hospital (Other)
Collaborators: Northeastern University (Other)
Responsible Party: Principal Investigator, Linda Bulich, Attending Anesthesiologist, Boston Children's Hospital
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: P00035987
Record Dates: First submitted 2020-09-15; First posted 2020-10-14 (Actual); Results first posted 2025-11-04 (Actual); Last update posted 2025-11-04 (Actual); Status verified 2025-10

CONDITIONS: Anesthesia; Anesthesia Emergence Delirium; Procedural Anxiety
Keywords: education
MeSH Terms: conditions — Emergence Delirium

STUDY DESIGN:
Who Masked: Care Provider, Outcomes Assessor
Masking Description: The research team member handing out surveys and observing children for anxiety are masked. The PACU nurse observing for emergence agitation post-op is also masked.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Standard Education (No Intervention): This group will receive the standard of care pre-operative education that all children get prior to ORL surgery at BCH Waltham.
- Pediatric Interactive Relational Agent (PIRA) (Experimental): This group will receive the standard of care pre-operative education that all children get prior to ORL surgery at BCH Waltham and will be given access to an interactive, online educational tool for use prior to surgery. This Pediatric Interactive Relational Agent (PIRA) will be able to be accessed as many times as the family would like prior to surgery.
  Interventions: Other: Pediatric Interactive Relational Agent (PIRA)

INTERVENTIONS:
Other: Pediatric Interactive Relational Agent (PIRA) — The PIRA is an interactive, online tool used to educate children and families about their child's upcoming surgical and anesthesia experience.
  Arms: Pediatric Interactive Relational Agent (PIRA)

SUMMARY:
The purpose of this study is to determine the efficacy of enhanced preoperative education using a Pediatric Interactive Relational Agent (PIRA), designed for children aged 4 through 10 years and their families, compared to the standard preoperative education currently provided. Specifically, the study aimed to evaluate differences in parent/child preoperative anxiety, and child experience with emergence from anesthesia. A secondary aim was to evaluate the child's and the parent's access and utilization the Pediatric Interactive Relational Agent as well as parental satisfaction and difficulties with the tool.

DETAILED DESCRIPTION:
This summary is a change from the original study/title where the secondary aim (from the original submission) is now the primary aim of the study and the primary aim (from the original submission) is now the secondary aim. This change was made following the first revision of the manuscript by the Editor in Chief and two separate reviewers. The manuscript was then rejected after a second review despite agreeing to reverse the primary and secondary outcomes as suggested by the reviewers. The Editor in Chief rejected this second submission stating that the newest revision (second revision) was not consistent with my original submission to ClinicalTrials.org. I am interested in submitting this manuscript to another journal yet wanted the changes to be updated in ClinicalTrials.org before resubmission.

ELIGIBILITY:
Inclusion Criteria:

* Parents (age 18+) and their children, ages 4 through 10 years old, who are undergoing general anesthesia and elective, outpatient ORL surgery at BCH Waltham
* American Society of Anesthesiology (ASA) physical status I or II
* Both parents and their children must be fluent in English

Exclusion Criteria:

* Parents without reliable internet access through a tablet or computer
* Parents of children with diagnosed developmental delays
* Parents who have children who have had previous surgical history under general anesthesia
* Parents of children involved in other anesthesia-related studies at BCH

Ages: 4 Years to 10 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 76 (Actual)
Dates: Start 2021-07-06 (Actual); Primary Completion 2023-10-19 (Actual); Study Completion 2023-10-19 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Linda Bulich, Principal Investigator — Boston Children's Hospital
Locations (1):
- Boston Children's Hospital, Waltham, Massachusetts, United States

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Standard Education | Pediatric Interactive Relational Agent (PIRA)
Started | 38 (number of parent/child dyads (i.e. 38 children and 38 parents/guardians)) | 38 (number of parent/child dyads (i.e. 38 children and 38 parents/guardians))
Completed | 35 (number of parent/child dyads (i.e. 35 children and 35 parents/guardians)) | 33 (number of parent/child dyads (i.e. 33 children and 33 parents/guardians))
Not Completed | 3 | 5
Not completed — Withdrawal by Subject | 0 | 2
Not completed — No longer eligible | 2 | 3
Not completed — Physician Decision | 1 | 0

BASELINE CHARACTERISTICS:
Population: Overall number of baseline participants refers to parent/guardian-child dyads. Baseline Measure Information (Age, Sex, Race/Ethnicity, etc) was not collected on the child participants.
Groups:
- Total: Total of all reporting groups
Arm/Group | Standard Education | Pediatric Interactive Relational Agent (PIRA) | Total
Number analyzed (Participants) | 38 | 38 | 76
Age, Continuous [Median (Inter-Quartile Range); unit: years] — Parental Age Population: In the Standard Education group, missing data is due to 3 dyads being withdrawn from the study due to surgery cancellation, research staff unavailability, inconsistent communication from parent, and 1 because the parent did not answer the age question on the survey.
  In the PIRA group, missing data is due to 4 dyads being withdrawn from the study due to the same reasons as above, and 2 parents did not answer the question on the survey.
  years
    number analyzed (Participants) | 34 | 32 | 66
    (all) | 40 [32 to 42] | 38 [34 to 39] | 38 [34 to 41]
Sex: Female, Male [Count of Participants; unit: Participants] — Parental sex Population: In the Standard Education group, missing data is due to 3 dyads being withdrawn from the study.
  In the PIRA group, missing data is due to 4 dyads being withdrawn from the study and 1 parent did not answer the sex question on the survey.
  Participants
    number analyzed (Participants) | 35 | 33 | 68
    Female | 31 | 32 | 63
    Male | 4 | 1 | 5
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants] — Parental Ethnicity Population: In the Standard Education group, missing data is due to 3 dyads being withdrawn from the study.
  In the PIRA group, missing data is due to 4 dyads being withdrawn from the study and 1 parent did not answer the ethnicity question on the survey.
  Participants
    number analyzed (Participants) | 35 | 33 | 68
    Hispanic or Latino | 1 | 1 | 2
    Not Hispanic or Latino | 31 | 32 | 63
    Unknown or Not Reported | 3 | 0 | 3
Race (NIH/OMB) [Count of Participants; unit: Participants] — Parental Race Population: In the Standard Education group, missing data is due to 3 dyads being withdrawn from the study prior to survey completion.
  In the PIRA group, 4 dyads were withdrawn from the study prior to survey completion and 1 parent did not answer the Race question.
  Participants
    number analyzed (Participants) | 35 | 33 | 68
    American Indian or Alaska Native | 0 | 0 | 0
    Asian | 0 | 1 | 1
    Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
    Black or African American | 1 | 3 | 4
    White | 31 | 28 | 59
    More than one race | 3 | 0 | 3
    Unknown or Not Reported | 0 | 1 | 1
Education Level of Parent/Guardian [Count of Participants; unit: Participants] — Population: In the Standard Education group, missing data is due to 3 dyads being withdrawn from the study prior to survey completion.
  In the PIRA group, 4 dyads were withdrawn from the study prior to survey completion and 1 parent did not answer the education question.
  Participants
    number analyzed (Participants) | 35 | 33 | 68
    Did Not Graduate High School | 0 | 0 | 0
    High School Diploma | 4 | 1 | 5
    Associate's Degree | 3 | 4 | 7
    Bachelor's Degree | 9 | 12 | 21
    Master's Degree | 12 | 15 | 27
    Doctoral Degree | 7 | 1 | 8

OUTCOME MEASURES:

1. Primary Outcome: Child Anxiety in Preoperative Waiting Room Using the Modified Yale Preoperative Anxiety Scale (mYPAS) for Child Anxiety
Description: The observational tool will be used to determine if there is a difference in anxiety between children who reviewed the PIRA and those who did not (control group). It will look at the incidence and severity of anxiety in children who received the PIRA vs. those who received standard preoperative education. This scale produces a score ranging from 22.92 to 100, with higher values indicating greater anxiety.
Time Frame: Preoperative Period - 1 day
Measure: Median (Inter-Quartile Range); unit: score on a scale
Arm/Group | Standard Education | Pediatric Interactive Relational Agent (PIRA)
Number analyzed (Participants) | 35 | 34
score on a scale | 25 [25 to 31.3] | 25 [25 to 25]

2. Primary Outcome: Parental Anxiety in Preoperative Waiting Room Using the Parental State-Trait Anxiety Inventory (STAI) for Parental Anxiety
Description: This survey will be used to determine if there a difference in anxiety between the parents who got the PIRA and those in the control group. It will look at the incidence and severity of anxiety in families who received the PIRA vs. those that received the standard education. Parental anxiety was assessed using the State-Trait Anxiety Inventory. The self-report anxiety instrument includes two separate 20-item subscales that measure trait (baseline) and state (situational) anxiety. The State-Trait Anxiety Inventory is scored from 20-80, with higher scores indicating more anxiety
Time Frame: Preoperative period- 1 day
Measure: Median (Inter-Quartile Range); unit: score on a scale
Arm/Group | Standard Education | Pediatric Interactive Relational Agent (PIRA)
Number analyzed (Participants) | 35 | 33
score on a scale | 46 [42 to 50] | 48 [43 to 50]

3. Primary Outcome: Emergence From Anesthesia: Presence or Absence of Emergence Agitation/Delirium (ED) Using the PACU Pediatric Anesthesia Emergence Delirium (PAED) for Anesthesia Scale
Description: This observational tool is used to determine if there is any effect on the incidence of emergence delirium for children who have more interactive preoperative education, such as PIRA, compared to standard information. The Post Anesthesia Emergence Delirium scale measures five behaviors, each rated on a five-point scale of 0 to 4. The scores are summed for a total score, with a maximum value of 20. An assessment of the internal consistency and reliability of the Post Anesthesia Emergence Delirium scale validated it for assessing emergence delirium in children recovering from general anesthesia.20 A score of >12 yields 100 percent sensitivity and 94.5 percent specificity for the diagnosis of emergence delirium. For this study, emergence delirium was considered present with a score of >12.
Time Frame: immediately postop in the PACU - 1 day
Measure: Median (Inter-Quartile Range); unit: score on a scale
Arm/Group | Standard Education | Pediatric Interactive Relational Agent (PIRA)
Number analyzed (Participants) | 35 | 33
score on a scale | 3 [0 to 10] | 4 [0 to 7]

4. Secondary Outcome: Parental Perceived Impact and Impressions Assessed Through the Parental PIRA Survey
Description: This survey assesses parental opinions about the PIRA.
Time Frame: Preoperative period - 1 day
Reporting Status: Not Posted

5. Secondary Outcome: Parental Utilization
Description: Interested in whether or not parents use the PIRA, frequency and duration of use and whether or not there were any barriers to its use. This will be assessed through the Parental PIRA survey.
Time Frame: 2-10 days before the day of surgery
Reporting Status: Not Posted

ADVERSE EVENTS:
Time Frame: Adverse even data were collected for length of time participants were in the study, which was up to 10 days.
Description: No adverse events were anticipated as this was a minimal risk study. As such, no adverse events occurred (all recorded deaths and adverse events are currently reported, as below). Adverse event reporting is for the parent/child dyad. The child participants in both groups were observed for preop anxiety and postop emergence delirium yet were not included in other arms of the study and were considered the same dyad with the parent/guardian.
Arm/Group | Standard Education | Pediatric Interactive Relational Agent (PIRA)
All-Cause Mortality (participants affected / at risk) | 0/35 | 0/34
Serious Adverse Events (participants affected / at risk) | 0/35 | 0/34
Other Adverse Events (participants affected / at risk) | 0/35 | 0/34

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2022-01-26): https://cdn.clinicaltrials.gov/large-docs/69/NCT04586569/Prot_SAP_000.pdf